CLINICAL TRIAL: NCT07042490
Title: Efficacy and Safety of Plasma Adsorption Combined With Endovascular Thrombectomy for Acute Ischemic Stroke Due to Large Vessel Occlusion of Anterior Circulation: A Multicenter, Randomized, Parallel-controlled Clinical Trial
Brief Title: Efficacy and Safety of Plasma Adsorption Combined With EVT for AIS-LVO
Acronym: PROMOTE-EVT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROMOTE-EVT
Record Dates: First submitted 2025-06-17; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-11

CONDITIONS: Acute Ischemic Stroke From Large Vessel Occlusion; Endovascular Thrombectomy
Keywords: Acute ischemic stroke; Plasma adsorption; Endovascular Thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Plasmapheresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma adsorption+Endovascular Thrombectomy (Experimental): Patients are received plasma adsorption and endovascular thrombectomy.Plasma adsorption was initiated after endovascular thrombectomy once daily for 3 days.
  Interventions: Procedure: Plasma adsorption; Procedure: Endovascular Thrombectomy
- Endovascular Thrombectomy (Active Comparator): The patients will be treated with endovascular thrombectomy .
  Interventions: Procedure: Endovascular Thrombectomy

INTERVENTIONS:
Procedure: Plasma adsorption — Plasma adsorption was initiated after endovascular thrombectomy once daily for 3 days.
  Arms: Plasma adsorption+Endovascular Thrombectomy
Procedure: Endovascular Thrombectomy — The patients will be treated with endovascular thrombectomy.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of plasma adsorption for patients of acute ischemic stroke who underwent endovascular thrombectomy due to large vessel occlusion of anterior circulation.

DETAILED DESCRIPTION:
Large vessel occlusive (LVO) stroke has a higher mortality and disability rate than other types of acute ischemic stroke (AIS). Endovascular thrombectomy (EVT) is recommended as a standard treatment for AIS-LVO. However, even if the blood vessels are successfully recanalization, nearly one-third of the patients still die and nearly half remain disabled at 3 months. Inflammation plays a crucial role in the pathophysiological cascade of ischemic stroke and related forms of brain injury. Evidence from experimental stroke indicates that targeting cytokines may reduce infarct volume and promote functional recovery. Plasma adsorption (PA) has been applied in the treatment of severe inflammatory diseases, including pancreatitis and sepsis, as well as in the neurological autoimmune diseases, such as myasthenia gravis, multiple sclerosis, and autoimmune encephalitis. We hypothesize that PA can improve functional outcome of AIS-LVO who underwent EVT.

In this study, the experimental group receive EVT and PA, 1 time per day for 3 consecutive days. The control group receive EVT . Two groups will be followed up for 90 days to evaluate the efficacy and safety of PA for patients of AIS-LVO of anterior circulation, who achieve successful recanalization through EVT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, male or female.
2. Diagnosis of acute ischemic stroke within 12 hours of symptom onset, underwent endovascular thrombectomy (EVT) adhering to current guidelines for large vessel occlusion in the anterior circulation (confirmed by DSA as ICA,MCA-M1,MCA-M2,ACA-A1,ACA-A2 occlusion or tandem lesion) and achieve successful recanalization (mTICI grade 2b/3).
3. Baseline NIHSS after EVT ≥ 6 and ≤25 points.
4. Randomization and the first plasma adsorption can be initiated within 12 hours after EVT.
5. Pre-stroke mRS≤ 2 points.
6. Patient/legally family members have signed the Informed consent form.

Exclusion Criteria:

1. Imaging after EVT indicated malignant brain edema with midline shift or brain herniation and surgical treatment was planned.
2. Parenchymal hemorrhage type 1, or type 2 confirmed by CT.
3. Allergic to any ingredient of the plasma separator, the adsorption device, or the piping.
4. Contraindications to plasma adsorption, platelet count <60×10^9/L,white blood cell<4×10^9/L, uncontrolled hypertension with persistent systolic blood pressure ≥200 mmHg or diastolic blood pressure ≥110 mmHg, uncontrolled hypotension, systolic blood pressure <90 mmHg or diastolic blood pressure <60 mmHg.
5. Previous history of malignant tumors, autoimmune diseases or being treated with immunosuppressants, hormones, or tumor necrosis factor inhibitors.
6. Previous history of organic heart disease and NYHA Class III or IV.
7. Currently taking anticoagulant(dabigatran, rivaroxiban, warfarin, etc.), previous history of serious hematological system disorders, or abnormal coagulation function (international normalized ratio [INR], activated partial thromboplastin time [APTT], prothrombin time [PT] upper limit of the normal range).
8. Severe liver and kidney dysfunction or abnormal laboratory test results（serum aspartate aminotransferase or alanine aminotransferase >3 times the upper limit of normal, serum creatinine>265umol/l(>3mg/dl)）.
9. Pregnancy , lactation or life expectancy of less than 3 months or inability to complete the study for other reasons.
10. Unwilling to be followed up or poor compliance.
11. Current or past participation in other clinical research, or participation in this study within 3 months prior to admission.
12. Other conditions that the researchers think make the patient unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) Score 0-2 at 90 days | 90±7 days
  Modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents a better outcome.

SECONDARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) Score 0-1 at 90 days | 90±7 days
  Modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents an excellent outcome.
Ordinal distribution of Modified Rankin Scale (mRS) | 90±7 days
  Modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death).
Proportion of patients with a reduction of NIHSS score（≥4 points） | 7 days(or discharge)
  The NIHSS is an ordinal hierarchical scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.
Blood lipid in peripheral blood | 72 hours, 7 days
  Blood lipid in peripheral blood，including total cholesterol, low-density lipoprotein cholesterol (LDL-C), and triglycerides. are assessed at 72 hours and 7 days from randomization.
Cytokine levels in peripheral blood | 72 hours, 7 days
  Cytokines such as pro-inflammatory factors including interleukins are assessed at 72 hours and 7 days from randomization.
Final infarct volume | 7 days (or discharge)
  Final infarct volume measured with diffusion weighted imaging (DWI) MRI.

OTHER OUTCOMES:
All-cause mortality | 90±7 days，at the discharge, whichever came first
  All-cause mortality is defined as death from any cause occurring during the study period.
Frequency of new intracerebral hemorrhage within 7 days | 7 days
  Evaluate new intracerebral hemorrhage， including symptomatic intracranial hemorrhage (sICH) and asymptomatic intracranial hemorrhage.
Frequency of adverse events within 90 days | 90±7 days
  Frequency of adverse events within 90 days.
Frequency of serious adverse events within 90 days | 90±7 days
  Frequency of serious adverse events within 90 days.
Frequency of adverse events associated with plasma adsorption within 90 days | 90±7 days
  Frequency of adverse events associated with plasma adsorption within 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenni Guo, MD,PhD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China